CLINICAL TRIAL: NCT01570478
Title: A 12-week, Multicenter, Randomized, Double-blind, Double-dummy, 2-arm Parallel Group Study Comparing the Efficacy and Safety of Foster® NEXThaler® (Beclomethasone Dipropionate 100 µg Plus Formoterol 6 µg/Actuation), 2 Inhalations b.i.d., Versus Seretide® Accuhaler® (Fluticasone 250 µg Plus Salmeterol 50 µg/Actuation), 1 Inhalation b.i.d., on Small Airway Derived Parameters in Patients With Asthma
Brief Title: A Study in Patients With Asthma
Acronym: NELSON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC/PR/15009/001/11; 2011-003449-17 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foster® NEXThaler® (Experimental): Foster® NEXThaler® (beclomethasone dipropionate 100 µg plus formoterol 6 µg per actuation), 2 inhalations b.i.d. (daily dose of BDP 400 µg plus FF 24 µg)
  Interventions: Drug: Foster® NEXThaler® 100/6 µg/unit dose
- Seretide® Accuhaler® (Active Comparator): Seretide® Accuhaler® (fluticasone propionate 250 μg plus salmeterol xinafoate 50 μg per actuation), 1 inhalation b.i.d. (daily dose of fluticasone 500 μg plus salmeterol 100 μg)
  Interventions: Drug: Seretide® Accuhaler® 250/50 µg/actuation

INTERVENTIONS:
Drug: Foster® NEXThaler® 100/6 µg/unit dose — Foster® NEXThaler® (beclomethasone dipropionate 100 µg plus formoterol 6 µg per actuation), 2 inhalations b.i.d. (daily dose of BDP 400 µg plus FF 24 µg)
  Arms: Foster® NEXThaler®
Drug: Seretide® Accuhaler® 250/50 µg/actuation — Seretide® Accuhaler® (fluticasone propionate 250 μg plus salmeterol xinafoate 50 μg per actuation), 1 inhalation b.i.d. (daily dose of fluticasone 500 μg plus salmeterol 100 μg)
  Arms: Seretide® Accuhaler®

SUMMARY:
The purpose of the present study is to demonstrate the higher efficacy of Foster® NEXThaler® 100/6 extra fine (two inhalations b.i.d.) versus Seretide® Accuhaler® 250/50 (one inhalation b.i.d.), in terms of pulmonary function (change from baseline to the end of treatment in post-dose peripheral airway resistance) in patients with asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease characterised by variable airflow obstruction and bronchial hyper responsiveness. Asthma affects both the large and the small airways and there is a growing body of evidence that small airways impairment is an important contributor to the pathogenesis and clinical expression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged ≥ 18, who have signed an Informed Consent form prior to initiation of any study-related procedure.
* Clinical diagnosis of asthma for a minimum of 12 months prior to screening confirmed by a chest physician according to international guidelines (GINA). The evidence of asthma must be confirmed through a documented (in the last three years) positive response to the reversibility test, defined as ΔFEV1 ≥ 12% and ≥ 200 mL over baseline, within 30 minutes after administration of 400 μg of salbutamol pMDI or through a documented (in the last three years) positive response to methacholine challenge test (PC20 < 8 mg/mL or PD20 < 1 mg).
* Baseline FEV1 > 80% of the predicted normal value after appropriate washout from bronchodilators (to be checked at screening and at randomisation visits).
* Asthma Control Test score ≥ 20 and < 25 (to be checked at screening and at randomisation visits).
* Impaired small airways function defined as baseline peripheral airway resistance [R(5Hz)-R(20Hz)] ≥ 0.07 kPa/L/s (to be checked at screening and at randomisation visits).
* Patients on previous regular treatment with Seretide® Accuhaler® (fluticasone propionate 250 μg plus salmeterol xinafoate 50 μg per actuation, daily dose of fluticasone 500 μg plus salmeterol 100 μg) at a stable dose for at least 2 months prior to inclusion.
* A cooperative attitude and ability to be trained to the proper use of DPI.

Main Exclusion Criteria:

* Patients with a diagnosis of COPD according to GOLD guidelines.
* Current smokers with a smoking history of > 10 pack/year.
* Patients who have a clinical or functional uncontrolled respiratory, haematological, immunologic, renal, neurologic, hepatic, endocrinal or other disease, or any condition that might, in the judgment of the investigator, represent for the patients an undue risk or that could compromise the results or interpretation of the study.
* History or current evidence of uncontrolled heart failure, clinically relevant coronary artery disease, recent myocardial infarction, severe hypertension, uncontrolled cardiac arrhythmias.
* Patients treated with LABA or ICS/LABA fixed combination in the 24 hours before the screening visit.
* Severe asthma exacerbation leading to intake of systemic corticosteroids (> 10 days) in the month before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatment in post-dose peripheral airway resistance [R(5Hz)-R(20Hz)]. | Baseline and 3 months

SECONDARY OUTCOMES:
Changes from baseline at each clinic visit in pre and post-dose Impulse Oscillometry (IOS)/plethysmographic/spirometric parameters | After 4, 8, 12 weeks of treatment
Asthma exacerbations (severe) | Up to 12 weeks of treatment
Clinical measures of asthma control | Up to 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Chetta, MD, Principal Investigator — Dept. of Cardiology and Pulmonary Medicine - Pama, Italy
Locations (1):
- Dipartimento Cardio-Polmonare - Azienda Ospedaliero-Universitaria - Padiglione Rasori, Parma, Italy

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-003449-17